CLINICAL TRIAL: NCT01951157
Title: A Randomized-Controlled Three-arm Phase II Study of Lurbinectedin (PM01183) Alone or In Combination With Gemcitabine and a Control Arm With Docetaxel as Second-Line Treatment in Unresectable Non-Small Cell Lung Cancer (NSCLC) Patients
Brief Title: A Clinical Study in Three-arm of Lurbinectedin (PM01183) Alone or in Combination With Gemcitabine and a Control Arm With Docetaxel as Second Line Treatment in Non-Small Cell Lung Cancer (NSCLC) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PM1183-B-004-13
Record Dates: First submitted 2013-09-17; First posted 2013-09-26 (Estimated); Results first posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Gemcitabine; PM 01183

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A - docetaxel (Active Comparator): 75 mg/m2 docetaxel day 1, 1-hour intravenous, every three weeks
  Interventions: Drug: Docetaxel
- B - lurbinectedin (PM01183) (Experimental): 3.2 mg/m2 PM01183, day 1, 1-hour intravenous, every three weeks
  Interventions: Drug: Lurbinectedin (PM01183)
- C - gemcitabine + lurbinectedin (PM01183) (Experimental): 800 mg/m2 gemcitabine / 1.6 mg/m2 PM01183 both on day 1 and day 8, 30-minutes gemcitabine/1-hour PM01183 intravenous, every three weeks
  Interventions: Drug: Gemcitabine; Drug: Lurbinectedin (PM01183)

INTERVENTIONS:
Drug: Docetaxel — Powder for solution for infusion
  Arms: A - docetaxel
Drug: Gemcitabine — Powder for solution for infusion
  Arms: C - gemcitabine + lurbinectedin (PM01183)
Drug: Lurbinectedin (PM01183) — Powder for concentrate for solution for infusion
  Arms: B - lurbinectedin (PM01183); C - gemcitabine + lurbinectedin (PM01183)

SUMMARY:
A clinical study of lurbinectedin(PM01183) alone or in combination with gemcitabine in comparison to docetaxel for the treatment of unresectable non-small cell lung cancer (NSCLC)patients

DETAILED DESCRIPTION:
A randomized-controlled, three-arm, phase II study of lurbinectedin (PM01183) alone or in combination with gemcitabine and a control arm with docetaxel as second-line treatment in unresectable non-small cell lung cancer (NSCLC)patients to evaluate the antitumor activity as progression-free survival at four months (PFS4) of PM01183 alone or in combination with gemcitabine as using single agent docetaxel as a reference in the control arm as current standard of care and to analyze overall survival (OS), overall survival rate at 1-year (OS12), duration of response (DR), antitumor activity, as response rate (RR), safety and efficacy profiles of PM01183 alone and in combination with gemcitabine, to be preliminary compared with docetaxel, patients' quality of life (QoL), pharmacokinetics (PK) of PM01183, pharmacokinetic/pharmacodynamic (PK/PD)correlation and pharmacogenomics (PGx)to explore potential correlations between clinical outcomes and molecular parameters found in tumor and blood samples

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed unresectable NSCLC
* Patients must have failed one prior line of CT-based therapy for unresectable disease
* Age between 18 and 75 years
* Eastern Cooperative Oncology Group (ECOG)performance status (PS) ≤ 1
* Adequate hematological, renal, metabolic and hepatic function
* At least three weeks since the last prior therapy, at least four weeks since completion of any prior radiotherapy
* Negative pregnancy test for pre-menopausal women

Exclusion Criteria:

* Concomitant diseases/conditions as unstable angina, myocardial infarction, symptomatic congestive heart failure or asymptomatic with left ventricular ejection fraction (LVEF) ≤ 50%, dyspnea, infection by human immunodeficiency virus (HIV), active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, active uncontrolled infection, pleural or pericardial effusions, myopathy, limitation of the patient's ability to comply with the treatment or to follow-up the protocol, any other major illness
* Histological features of neuroendocrine or bronchioalveolar differentiation.
* Unknown epidermal growth factor receptor (EGFR)mutation status or previously known EGFR mutated status in patients with adenocarcinoma.
* Prior or concurrent invasive malignant disease, unless in complete remission for more than three years.
* Significant cancer-related weight loss (≥10%)within four weeks prior to treatment start
* Prior treatment with docetaxel-containing therapy
* Symptomatic, steroid-requiring or progressive central nervous system (CNS) involvement
* Paraneoplastic syndromes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2013-09-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 69 patients were enrolled between 11/09/2013 and 2/10/2015 at 13 centers. 68 patients were treated: 22 in Arm A, 21 in Arm B, and 25 in Arm C. The first dose of the first cycle was administered on 17/09/2013 and the last dose of the last cycle was administered on 3/11/2016. The last patient, last follow-up was on 24/11/2016
Groups:
- B - Lurbinectedin (PM01183): In the first protocol version, PM01183 7 mg Flat dose, 1-h i.v. infusion (at a fixed rate), on D1, q3wk, up to 6 cycles After protocol amendment 3, PM01183 3.2 mg/m2, 1-h i.v. infusion (at a fixed rate), on D1, q3wk, up to 6 cycles
  Lurbinectedin (PM01183): Powder for concentrate for solution for infusion
- C - Gemcitabine + Lurbinectedin (PM01183): Gemcitabine 800 mg/m2, 30-min i.v. infusion, immediately followed by PM01183 3.0 mg Flat dose, 1-h i.v. infusion (at a fixed rate), on D1, q3wk, up to 6 cycles (in the first protocol version) or PM01183 1.6 mg/m2, 1-h i.v. infusion (at a fixed rate), on D1, q3wk, up to 6 cycles (after protocol amendment 3)
  Gemcitabine: Powder for solution for infusion
  Lurbinectedin (PM01183): Powder for concentrate for solution for infusion
Period: Overall Study
Arm/Group | A - Docetaxel | B - Lurbinectedin (PM01183) | C - Gemcitabine + Lurbinectedin (PM01183)
Started | 22 | 22 | 25
Completed | 0 | 0 | 0
Not Completed | 22 | 22 | 25
Not completed — Progressive Disease | 12 | 13 | 10
Not completed — Treatment-unrelated AE | 1 | 0 | 3
Not completed — Study Termination | 0 | 0 | 1
Not completed — Physician Decision | 5 | 3 | 2
Not completed — Non-treatmentrelated death | 2 | 2 | 2
Not completed — No treated | 0 | 1 | 0
Not completed — Treatment-related AE | 2 | 0 | 4
Not completed — Consent withdrawn by subject | 0 | 1 | 3
Not completed — Treatment-related death | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: 69 patients were enrolled between 11/09/2013 and 2/10/2015 at 13 centers. 68 patients were treated: 22 in Arm A, 21 in Arm B, and 25 in Arm C. The first dose of the first cycle was administered on 17/09/2013 and the last dose of the last cycle was administered on 3/11/2016. The last patient, last follow-up was on 24/11/2016
Groups:
- Total: Total of all reporting groups
Arm/Group | A - Docetaxel | B - Lurbinectedin (PM01183) | C - Gemcitabine + Lurbinectedin (PM01183) | Total
Number analyzed (Participants) | 22 | 22 | 25 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 10 | 13 | 38
  >=65 years | 7 | 12 | 12 | 31
Age, Continuous [Median (Full Range); unit: years] | 61.5 [49 to 72] | 65 [46 to 74] | 64 [41 to 75] | 63 [41 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 9 | 19
  Male | 17 | 17 | 16 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 21 | 22 | 25 | 68
  Race: Unknown | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 0 | 0 | 2
  Italy | 8 | 11 | 13 | 32
  Belgium | 0 | 3 | 0 | 3
  Spain | 12 | 8 | 12 | 32
ECOG PS [Count of Participants; unit: Participants] — ECOG PS, Eastern Cooperative Oncology Group performance status PS 0 Fully active, able to carry on all pre-disease performance without restriction PS 1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature PS 2 Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours PS 3 Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours PS 4 Completely disabled; cannot carry on any selfcare; totally confined to bed or chair PS 5 Dead
  Participants
    PS 0 | 6 | 11 | 10 | 27
    PS 1 | 16 | 11 | 15 | 42
Histology type [Count of Participants; unit: Participants]
  Non-squamous-cell | 17 | 18 | 19 | 54
  Squamous-cell | 4 | 4 | 6 | 14
  Not specified | 1 | 0 | 0 | 1
Histology grade [Count of Participants; unit: Participants]
  Well differentiated | 0 | 1 | 0 | 1
  Moderately differentiated | 2 | 5 | 1 | 8
  Poorly differentiated | 7 | 3 | 9 | 19
  Unknown | 13 | 13 | 15 | 41
Stage at diagnosis [Count of Participants; unit: Participants]
  Early | 1 | 1 | 2 | 4
  Locally advanced | 4 | 7 | 4 | 15
  Metastatic | 15 | 14 | 18 | 47
  Unknown | 2 | 0 | 1 | 3
Stage at study entry [Count of Participants; unit: Participants]
  Locally advanced | 1 | 0 | 2 | 3
  Metastatic | 21 | 22 | 23 | 66
Surgery [Count of Participants; unit: Participants]
  Yes | 3 | 5 | 3 | 11
  No | 19 | 17 | 22 | 58
Radiotherapy [Count of Participants; unit: Participants]
  Yes | 9 | 10 | 10 | 29
  No | 13 | 12 | 15 | 40
Prior chemotherapy [Count of Participants; unit: Participants] — Number of prior lines
  Participants
    1 line | 19 | 21 | 23 | 63
    2 lines | 3 | 1 | 2 | 6
Best response to last prior platinum [Count of Participants; unit: Participants] — Best response to last prior platinum based chemotherapy NA, not applicable; PD, progressive disease; PR, partial response; SD, stable disease; UK, unknown
  Participants
    PR | 11 | 11 | 9 | 31
    SD | 5 | 8 | 10 | 23
    PD | 5 | 3 | 5 | 13
    NA | 1 | 0 | 0 | 1
    UK | 0 | 0 | 1 | 1
Weight [Median (Full Range); unit: Kg] | 70.5 [45 to 90.8] | 74 [39 to 124] | 77 [40 to 136] | 73.6 [39 to 136]
Body Surface Area [Median (Full Range); unit: m^2] | 1.8 [1.4 to 2.1] | 1.9 [1.4 to 2.3] | 1.9 [1.3 to 2.5] | 1.8 [1.3 to 2.5]
Signs and symptoms per patient [Median (Full Range); unit: Signs and symptoms] — Prior history per patient by MedDRA category, eg., cough, dyspnea, fatigue...
  Signs and symptoms | 1 [0 to 4] | 1 [0 to 4] | 1 [0 to 5] | 1 [0 to 5]
Albumin [Median (Full Range); unit: g/dL] | 4.3 [3.1 to 4.7] | 3.9 [3.2 to 5] | 4 [3.3 to 4.8] | 4 [3.1 to 5]
Alpha-1-acid glycoprotein [Median (Full Range); unit: mg/dL] | 172 [144 to 251] | 141 [65 to 243] | 159 [57 to 247] | 161 [57 to 251]
Time from first diagnosis to first infusion [Median (Full Range); unit: months] | 8 [2.4 to 48] | 11.4 [3.3 to 42.7] | 9.2 [1.9 to 109.3] | 9.8 [1.9 to 109.3]
Number of sites involved at baseline [Median (Full Range); unit: sites] | 3 [1 to 6] | 3 [1 to 6] | 3 [1 to 6] | 3 [1 to 6]
Platinum-free interval [Median (Full Range); unit: months] | 3.5 [1 to 16.3] | 5.6 [0.7 to 36.8] | 3.9 [1 to 20.8] | 4.4 [0.7 to 36.8]
PFS to last prior line [Median (Full Range); unit: mohths] — PFS, progression-free survival Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression
  mohths | 5.7 [0.1 to 18.2] | 6.7 [1.1 to 36.9] | 5.4 [1.1 to 17.4] | 5.8 [0.1 to 36.9]

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Rate at Four Months (PFS4)
Description: The rate estimate of the percentage of patients who are alive and progression-free at 16 weeks (~4 months) after randomization. Progession disease was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression.
Time Frame: At month four after patient inclusion
Population: Arm B: 1 no treated, 1 no tumour assesment, 1 major protocol deviation Arm C: 2 no tumour assesment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A - Docetaxel | B - Lurbinectedin (PM01183) | C - Gemcitabine + Lurbinectedin (PM01183)
Number analyzed (Participants) | 22 | 19 | 23
percentage of participants | 27.3 [10.7 to 50.2] | 15.8 [3.4 to 39.6] | 26.1 [10.2 to 48.4]
Statistical Analysis 1: Comparison: A - Docetaxel; The exact binomial estimator and its 95%CI was used. A pre-planned Bayesian supportive analysis test comparing PFS4 was performed; Test type: Superiority; The exact binomial estimator = 29.2, 95% CI 2-sided [13.2 to 48.4]
Statistical Analysis 2: Comparison: B - Lurbinectedin (PM01183); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; The exact binomial estimator = 19.0, 95% CI 2-sided [5.7 to 37.9]
Statistical Analysis 3: Comparison: C - Gemcitabine + Lurbinectedin (PM01183); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; The exact binomial estimator = 28.0, 95% CI 2-sided [12.6 to 46.7]

2. Secondary Outcome: Progression-free Survival
Description: PFS, progression-free survival Progression-free survival (PFS), defined as the time from the date of randomization to the date of PD, death (of any cause), or last tumor evaluation. Progession disease was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression.
Time Frame: Time from the date of randomization to the date of PD, death (of any cause), or last tumor evaluation, whichever came first, assessed up to 3 years
Population: B- 1 no treated, 1 no tumour assesment, 1 major protocol deviation C - 2 no tumour assesment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A - Docetaxel | B - Lurbinectedin (PM01183) | C - Gemcitabine + Lurbinectedin (PM01183)
Number analyzed (Participants) | 22 | 19 | 23
months | 3.1 [1.8 to 4] | 1.9 [1.5 to 3] | 3.3 [1.9 to 5.7]
Statistical Analysis 1: Comparison: A - Docetaxel vs B - Lurbinectedin (PM01183) vs C - Gemcitabine + Lurbinectedin (PM01183); Test type: Superiority — Pre-specified; p = 0.3873, Log Rank

3. Secondary Outcome: Progression-free Survival Rate at Six Months (PFS6)
Description: The rate estimate of the percentage of patients who are alive and progression-free at 24 weeks (~6 months) after randomization. Progession disease was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression.
Time Frame: At month six after patient inclusion
Population: B- 1 no treated, 1 no tumour assesment, 1 major protocol deviation C - 2 no tumour assesment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A - Docetaxel | B - Lurbinectedin (PM01183) | C - Gemcitabine + Lurbinectedin (PM01183)
Number analyzed (Participants) | 22 | 19 | 23
percentage of participants | 18.2 [2.1 to 34.3] | 16.7 [0 to 33.9] | 17.5 [0 to 35.2]

4. Secondary Outcome: Overall Response Rate
Description: Overall response rate (ORR) was defined as the percentage of patients with a response, either CR or PR, according to RECIST v.1.1.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Time from the date of randomization until 30±7 days after the last treatment infusion, assessed up to 3 years
Population: B - 1 no treated, 1 no tumour assesment, 1 major protocol deviation C - 2 no tumour assesment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A - Docetaxel | B - Lurbinectedin (PM01183) | C - Gemcitabine + Lurbinectedin (PM01183)
Number analyzed (Participants) | 22 | 19 | 23
percentage of participants | 9.1 [1.1 to 29.2] | 0 [0 to 17.6] | 17.4 [5.0 to 38.8]

5. Secondary Outcome: Objective Response Per RECIST v.1.1
Description: RECIST, Response Evaluation Criteria In Solid Tumors Complete Response (CR) Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10mm Partial Response (PR) At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters Progressive Disease (PD) At least a 20% increase in the sum of diameters of target lesions taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. Appearance of new lesions was considered PD Stable Disease (SD) Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as reference the smallest sum diameters while on study Treatment failure (TF) Symptomatic deterioration/death due to progression or treatment discontinuation due to treatment-related toxicity occurred before any appropriate tumor assessments had been performed
Time Frame: Time from the date of randomization until 30±7 days after the last treatment infusion, assessed up to 3 years
Population: B- 1 no treated, 1 no tumour assesment, 1 major protocol deviation C- 2 no tumour assesment
Measure: Count of Participants; unit: Participants
Arm/Group | A - Docetaxel | B - Lurbinectedin (PM01183) | C - Gemcitabine + Lurbinectedin (PM01183)
Number analyzed (Participants) | 22 | 19 | 23
Participants
  PR | 2 | 0 | 4
  SD | 10 | 7 | 11
  PD | 8 | 8 | 6
  TF | 2 | 4 | 2

6. Secondary Outcome: Duration of Response
Description: Duration of response (DR) was defined as the time from the date when the response criteria (PR or CR, whichever was reached first) were fulfilled, to the first date when PD, recurrence or death was documented.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: The time from the date when the response criteria (PR or CR, whichever was reached first) were fulfilled, to the first date when PD, recurrence or death was documented, up to 3 years
Population: Two patients with CR or PR to treatment as per the RECIST v.1.1 criteria were found in Arm A.
  No patients with CR or PR to treatment as per the RECIST v.1.1 criteria were found in Arm B.
  Four patients with CR or PR to treatment as per the RECIST v.1.1 criteria were found in Arm C.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A - Docetaxel | B - Lurbinectedin (PM01183) | C - Gemcitabine + Lurbinectedin (PM01183)
Number analyzed (Participants) | 2 | 0 | 4
months | 1.2 [0.8 to 1.6] |  | 6.1 [2.0 to NA] — upper limit was not estimable due to few participants with events
Statistical Analysis 1: Comparison: A - Docetaxel vs C - Gemcitabine + Lurbinectedin (PM01183); Test type: Superiority — Pre-specified; p = 0.0177, Log Rank

7. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) will be defined as time from the date of first infusion to the date of death or last contact
Time Frame: From the date of first infusion to the date of death or last contact, up to 12 months after last patient inclusion
Population: Arm B: 1 no treated, 1 no tumour assesment, 1 major protocol deviation Arm C: 2 no tumour assesment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A - Docetaxel | B - Lurbinectedin (PM01183) | C - Gemcitabine + Lurbinectedin (PM01183)
Number analyzed (Participants) | 22 | 19 | 23
months | 9.4 [3.1 to NA] — upper limit was not estimable due to few participants with events | 5.5 [3.0 to 8.0] | 7.2 [4.5 to 10.6]
Statistical Analysis 1: Comparison: A - Docetaxel vs B - Lurbinectedin (PM01183) vs C - Gemcitabine + Lurbinectedin (PM01183); Test type: Superiority or Other — Pre-specified; p = 0.3526, Log Rank

8. Secondary Outcome: Information on Quality of Life (QoL)
Description: The mean QoL scores self-reported by patients using the Lung Cancer Symptom Scale (LCSS) at baseline and after the start of the therapy in visits 3 or 6 (+/- 1 visit) and visit 9 for those patients in maintenance therapy.
  Higher LCSS scores indicate more severe problems and the scale range is (0-100) Total score was calculated as the mean of the total scores of all nine patient ítems (Appetite, Fatigue, Cough, Dyspnea, Hemoptysis, Pain, Lung cancer symptoms, Normal activities, Global QoL)
Time Frame: Baseline, Cycle 3 (~9 weeks), Cycle 6 (~18 weeks) and Cycle 9 (~27 weeks)
Population: No patients in cycle 9 in arm A and arm C.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | A - Docetaxel | B - Lurbinectedin (PM01183) | C - Gemcitabine + Lurbinectedin (PM01183)
Number analyzed (Participants) | 22 | 20 | 25
units on a scale
  Baseline | 27.2 [18.4 to 36.1] | 36.4 [25.0 to 47.7] | 38.1 [27.7 to 48.5]
  Cycle 3: number analyzed (Participants) | 11 | 10 | 12
  Cycle 3 | 29.5 [14.5 to 44.5] | 32.2 [19.5 to 44.9] | 36.4 [25.4 to 47.5]
  Cycle 6: number analyzed (Participants) | 5 | 1 | 3
  Cycle 6 | 24.3 [17.4 to 31.1] | 55.4 [NA to NA] — 95%CI was not calculated due to only one patient was evaluated | 35.4 [-11.7 to 82.5]
  Cycle 9: number analyzed (Participants) | 0 | 2 | 0
  Cycle 9 |  | 38.1 [-74.8 to 151.1] |
Statistical Analysis 1: Comparison: A - Docetaxel; Changes in QoL scores over time were calculated and tested for statistical significance by means of wilcoxon signed ranks test repeat-measure analyses of variance; Test type: Superiority — Pre-specified; p = 0.9026, Wilcoxon signed ranks test repeat analys
Statistical Analysis 2: Comparison: B - Lurbinectedin (PM01183); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.9862, Wilcoxon signed ranks test repeat analys
Statistical Analysis 3: Comparison: C - Gemcitabine + Lurbinectedin (PM01183); Changes in QoL scores over time were calculated and tested for statistical significance by means of ilcoxon signed ranks test repeat-measure analyses of variance; Test type: Superiority; p = 0.8057, Wilcoxon signed ranks test repeat analys

ADVERSE EVENTS:
Time Frame: Participants were assessed through study completion, approximately 3 years
Description: All 68 treated patients were evaluable for safety: 22 in Arm A (docetaxel), 21 in Arm B (PM01183) and 25 in Arm C (gemcitabine/PM01183). One Patient in Arm B was never treated due to patient's refusal, therefore, this patient was excluded of the safety population
Groups:
- B - Lurbinectedin (PM01183): In the first protocol version, PM01183 7 mg Flat dose, 1-h i.v. infusion (at a fixed rate), on D1, q3wk, up to 6 cycles After protocol amedment 3, PM01183 3.2 mg/m2, 1-h i.v. infusion (at a fixed rate), on D1, q3wk, up to 6 cycles
  Lurbinectedin (PM01183): Powder for concentrate for solution for infusion
- C - Gemcitabine + Lurbinectedin (PM01183): Gemcitabine 800 mg/m2, 30-min i.v. infusion, immediately followed by PM01183 3.0 mg Flat dose, 1-h i.v. infusion (at a fixed rate), on D1, q3wk, up to 6 cycles (in the first protocol version) or PM01183 1.6 mg/m2, 1-h i.v. infusion (at a fixed rate), on D1, q3wk, up to 6 cycles (after protocol amedment 3)
  Gemcitabine: Powder for solution for infusion
  Lurbinectedin (PM01183): Powder for concentrate for solution for infusion
Arm/Group | A - Docetaxel | B - Lurbinectedin (PM01183) | C - Gemcitabine + Lurbinectedin (PM01183)
All-Cause Mortality (participants affected / at risk) | 14/22 | 17/21 | 21/25
Serious Adverse Events (participants affected / at risk) | 12/22 | 9/21 | 18/25
Other Adverse Events (participants affected / at risk) | 21/22 | 20/21 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A - Docetaxel (N=22) | B - Lurbinectedin (PM01183) (N=21) | C - Gemcitabine + Lurbinectedin (PM01183) (N=25)
Shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia/Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 2 (8) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (3) | 1 (1) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 3 (4)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0) | 4 (4)
Septic shock (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Candida pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A - Docetaxel (N=22) | B - Lurbinectedin (PM01183) (N=21) | C - Gemcitabine + Lurbinectedin (PM01183) (N=25)
Phlebitis (Vascular disorders) | 0 (0) | 1 (6) | 2 (3)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (3)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Asthenia/Fatigue (General disorders) | 16 (30) | 16 (32) | 17 (35)
Mucosal inflammation (General disorders) | 4 (4) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 4 (5) | 2 (3) | 5 (7)
Pyrexia (General disorders) | 7 (10) | 5 (8) | 7 (14)
Chest pain (General disorders) | 0 (0) | 2 (2) | 3 (3)
General physical health deterioration (General disorders) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 2 (4) | 3 (6)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 4 (5)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 7 (11) | 15 (29)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 3 (8) | 13 (21)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (13) | 5 (7) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 5 (7) | 7 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 4 (4) | 1 (1) | 2 (5)
Conjunctivitis (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 5 (6) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 3 (5) | 3 (4) | 4 (10)
Nausea (Gastrointestinal disorders) | 2 (2) | 6 (7) | 13 (23)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (4)
Vomiting (Gastrointestinal disorders) | 2 (4) | 8 (10) | 6 (13)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 6 (7) | 3 (4)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (5) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (4) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (6) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 10 (13) | 8 (10)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 3 (3) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (3) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review